CLINICAL TRIAL: NCT05128656
Title: Kinetic of Humoral Immune Response of Asymptomatic Nursing Homes (EHPAD) Employees Infected With Severe Acute Respiratory Syndrome Coronavirus : a Case Control Study
Brief Title: Immune Response of Asymptomatic EHPAD Employees Infected With COVID-19
Acronym: SERASYMPTO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Authorization denied by Ethical Comitee
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: APHP201253; 2020-A01833-36 (Other: ID-RCB)
Record Dates: First submitted 2020-11-19; First posted 2021-11-22 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
Keywords: EHPAD employees; COVID-19; asymptomatic; humoral response
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Case control longitudinal study, Interventional minimal risk study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cases (Other): SARS-Cov-2 asymptomatic nursing homes employees
  Interventions: Other: serology
- Controls (Other): cohort of patients with a symptomatic COVID-19, preferably recruited in nursing homes or in case of difficulties in the virology service of COCHIN Hospital.
  Interventions: Other: serology

INTERVENTIONS:
Other: serology — serology at M3 and serology at M6

SUMMARY:
The investigators performed in April 2020, a screening campaign of asymptomatic staff working in elderly nursing homes in Paris France (EHPAD), where the virus had been circulating actively in March and April 2020. Among 241 employees tested in four nursing homes, 32 (13.2%) were asymptomatic carriers of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-Cov-2).

Few data are available concerning the humoral immune response of asymptomatic carriers, the elicitation and duration of neutralizing antibodies and the duration of protection.

The purpose of the study is to determine whether these asymptomatic persons develop a humoral immune response, whether this immune response is durable and whether it is protective against the risk of reinfection

DETAILED DESCRIPTION:
The investigators performed in April 2020, a screening campaign of asymptomatic staff working in elderly nursing homes in Paris, France, where the virus had been circulating actively in March and April 2020. Among 241 employees tested in four nursing homes, 32 (13.2%) were asymptomatic carriers of SARS-Cov-2.

Few data are available concerning the humoral immune response of asymptomatic carriers, the elicitation and duration of neutralizing antibodies and the duration of protection.

The main objective of this study is to describe the SARS-Cov-2 asymptomatic employees with positive immunoglobulin G (igG) serology at month 1-2 post infection.

Secondary objectives are

* To describe the proportion of asymptomatic persons with SARS-Cov-2 antibodies month 3 and 6 post infection
* To compare the proportion of persons with SARS-Cov-2 antibodies between asymptomatic and asymptomatic carriers at M1-2 post infection, M3 and M6 post infection
* To determine the factors associated with the appearance of antibodies ( viral load, age, sex, previous history, habitus..)
* To study the neutralizing capacities and immune-profiling of SARS-Cov-2 antibodies in vitro
* To evaluate the occurrence of Coronavirus Disease 2019 (COVID-19) reinfections in asymptomatic carriers during the second wave.

The design will be a case control study between

* Cases: SARS-Cov-2 asymptomatic nursing homes employees
* Controls: cohort of patients with a symptomatic COVID-19, preferably recruited in nursing homes or in case of difficulties in the virology service of COCHIN Hospital.

ELIGIBILITY:
* Common inclusion criteria:

  * Age ≥ 18.
  * Health care employees working in the EHPAD who consulted in the Hotel Dieu Hospital
  * Affiliated with a health insurance
  * Informed information and consent
* Inclusion Criteria for Cases (asymptomatic COVID-19 patients) :

  * Health care workers screened SARS-Cov-2 positive for NASopharyngeal swaths during screening campaigns for EHPAD staff.
  * Having carried out a follow-up serology (M1 and M2) within the Hotel Dieu.
  * Having never developed symptoms of COVID-19 or have developed some symptoms undetected before screening: fever, transient fatigue, rhinorrhea, symptoms that may be mistaken for a common winter cold (no respiratory symptoms or prolonged fever)
* Inclusion criteria for controls (symptomatic COVID-19 patients) :

  * Health care workers tested positive for polymerase chain reaction assay (PCR) SARS-Cov-2 during screening campaigns for EHPAD staff at the Hotel Dieu.
  * Having carried out a follow-up serology (M1 and M2) within the Hotel Dieu.

COVID-19 symptoms defined by:

* At least two major signs of COVID-19 among: > fever, cough, chest tightness, bilateral pneumonia, anosmia, loss of taste.
* or a major sign and three minor signs among: headache, severe fatigue, diarrhea, odynophagia, rhinorrhea, suggestive skin signs.

It is part of the database of the virology department of Cochin Hospital (in case of failure to recruit health care workers in the EHPADs).

*Exclusion criteria :

* Refuse to participate or inability to obtain informed consent.
* under guardianship, curators
* negative SARS-COV-2 PCR
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-18 (Actual); Primary Completion 2022-06-18 (Actual); Study Completion 2022-06-18 (Actual)

PRIMARY OUTCOMES:
rate of positive IgG serology | month 1-2 post infection
  positive IgG (Immunoglobulin G) SARS-Cov-2 serology after infection of asymptomatic employees

SECONDARY OUTCOMES:
rate of positive IgG serology | month 3-6 post infection
  positive IgG (Immunoglobulin G) SARS-Cov-2 serology after infection of asymptomatic employees
rate of positive immunoglobulin M (IgM) serology | month 1-2-3 and 6 post infection
  positive IgM SARS-Cov-2 serology after infection of asymptomatic employees
rate of neutralizing antibodies | month 1-2-3 and 6 post infection
  concentration of neutralizing antibodies
questionnaire | month 1-2-3 and 6 post infection
  Associated factors with the presence of antibodies
re infection | through study completion, an average of 8 months
  of asymptomatic patients with SARS-Cov-2

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Salmon, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- HOTEL DIEU Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No